CLINICAL TRIAL: NCT02505009
Title: Efficacy of HBV Therapeutic Vaccine in Consolidation of Nucleos(t)Ide Analogues Therapy: a Pilot Study
Brief Title: Efficacy of HBV Vaccine in Consolidation of Nucleos(t)Ide Analogues Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 104-3167C
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2018-12

CONDITIONS: Chronic Hepatitis B
Keywords: Therapeutic Uses; Entecavir; Tenofovir; Engerix-B; DNA Virus Infections; Antiviral Agents; Vaccination
MeSH Terms: conditions — Hepatitis B, Chronic; DNA Virus Infections | interventions — Engerix-B; Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- entecavir pretreated vaccine arm (Experimental): Arm A,case group: 75 cases will be enrolled to receive Engerix-B injection and compared with histological non-vaccine treated controls
  Interventions: Drug: Engerix-B; Drug: Entecavir
- tenofovir pretreated vaccine arm (Experimental): Arm B case group: A total of 50 patients will be randomized into case (vaccine) and control group according to age, gender, pretreatment HBV DNA level.
  Interventions: Drug: Engerix-B; Drug: Tenofovir
- Entecavir pretreated control arm (Active Comparator): Arm A control group: Age, gender and pretreatment DNA matched histological controls
  Interventions: Drug: Entecavir
- tenofovir pretreated control arm (Active Comparator): Arm B control group: A total of 50 patients will be randomized into case (vaccine) and control group according to age, gender, pretreatment HBV DNA level.
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Engerix-B — The case group will receive 5 Engerix-B injections during the last 6 months of a 3-year NA therapy.
  Arms: entecavir pretreated vaccine arm; tenofovir pretreated vaccine arm
Drug: Tenofovir — Both case and control will receive 300 mg Tenofovir for at least 3 years
  Arms: tenofovir pretreated control arm; tenofovir pretreated vaccine arm
Drug: Entecavir — Both case and control will receive 0.5 mg entecavir therapy for at least 3 years
  Arms: Entecavir pretreated control arm; entecavir pretreated vaccine arm

SUMMARY:
Background and aims: Nucleos(t)ide analogues may suppress HBV DNA to undetectable level, but only about 30-40% remain sustained response 1-3 years after discontinued therapy. The investigators will try to improve the sustained response rate by given a course of HBV vaccination during the last 6 months on patients receiving a 3-year entecavir or tenofovir therapy.

Rational: The host may response to HBV vaccine when HBV DNA and immune tolerance are suppressed during entecavir or tenofovir therapy.

Patients: Patients who have been receiving entecavir or tenofovir therapy for at least 30 months will be invited to this study. The case group will receive 5 Engerix-B injections during the last 6 months of entecavir or tenofovir therapy. Arm A-entecavir pretreated group: 75 cases will be enrolled to receive Engerix-B injection and compared with histological non-vaccine treated controls; Arm B-tenofovir pretreated group: 50 patients will be randomized into case (vaccine) and control group according to age, gender, pretreatment HBV DNA level.

Therapy: Both case and control groups will receive a 3 year or longer entecavir or tenofovir therapy. Patients will be screen at 24-30 months and enrolled at 30 months after entecavir or tenofovir therapy. They will receive 5 Engerix-B injections at 0,1st ,2nd,3rd and 6th month [30-36 +/-1 month post nucleos(t)ide therapy] post enrollment. Both drugs will be discontinued after completed therapy.

Follow-up: Both groups will be monitoring by biochemistry, alpha-fetoprotein, quantitative HBsAg, HBV DNA levels and immunological parameter periodically for 2 years after therapy.

Efficacy: Those patients with persistent normal ALT and HBV DNA lower than 1*100000 cps/mL after discontinued nucleos(t)ide analogues therapy will be considered to have sustained response. Patients with transient elevation of HBV DNA and ALT, but normalized spontaneously without further therapy will be defined as delayed response. Patients with persistent HBV DNA greater than 1*100000 cps/mL will be considered to have non-sustained response.

Study duration: The enrollment will be completed in one year and keep on observation for additional 2 years.

Expected goals of the study: HBV vaccine and nucleos(t)ide analogues combination therapy may decrease the HBV relapse rate at 1 and 2 year after completed therapy.

DETAILED DESCRIPTION:
Introduction Chronic hepatitis B virus (HBV) infection is a widely prevalent global health problem with estimate 350-400 million chronic HBV carriers worldwide. In China, Southeast Asia and sub-Saharan Africa, as many as 10-15% of the population are chronically infected with HBV. In North America and North Europe, HBV chronic carrier rates are much lower, usually below 1%. Intermediate HBV carrier rates of 1-7% are found in parts of Southern and Eastern Europe, Central America, the Middle East and parts of Japan (1-4).

HBV is highly infectious; many chronic HBsAg carriers were infected in their family shortly after birth or in early childhood (5-7). Recent genome-wide association studies revealed antigen presenting molecules, Human leukocyte antigen-DP (HLA-DP) and HLA-DQ, are associated with persistence HBV infection (8-10). HBV is actively replicated in chronic carriers during the initial immune tolerance phase (11). Impaired innate and adaptive immune responses to HBV can be found during this stage (12-16). They are generally asymptomatic until the immune clearance phase developed. At this stage, innate immunity, HBV-specific and non-specific T cells and other immune cells may orchestra an immune response and hepatic necroinflammation to clear HBV (17-19). The immune clearance phase is critical to the outcome of chronic HBsAg carriers. Those patients with prolonged HBV replication and repeated hepatic inflammation will run into liver cirrhosis and /or hepatocellular carcinoma (HCC) (20-23). How to terminate HBV replication is an important issue in management of chronic HBsAg carriers.

1.1 Therapy for chronic hepatitis B In the past 20 years, significant improvements in treatment of chronic hepatitis B (CHB) have been achieved by introducing regimen of interferon derivatives and nucleotide/nucleoside analogues (NA) (24-26). Interferon is a T helper cell type 1 cytokine that promotes immunity of host to clear HBV (27,28). NA inhibit HBV DNA synthesis by termination the nascent proviral DNA chain. About 30% patients may have complete response with normalization alanine aminotransferase (ALT) and HBV DNA lower than 10000 cps/mL one to three year after discontinued therapy (10,29-31). For the rest of patients a flare-up HBV replication occurred (10,29-31), a life-long therapy may be needed to eliminate covalently closed circular DNA (cccDNA) pool and achieved a sustained therapeutic response (32). Unfortunately, the prolonged use of NA need a lot of budgets and carried a substantial risk for emerging drug resistance mutants (33). The interferon derivatives regimens have similar efficacy with significant side effects (27,28). Therefore, Development of a safe and affordable anti-HBV agent/strategy is needed to further improve outcomes (34).

1.2 Rational for combine HBV vaccine with NA therapy NA therapy may suppress Serum HBV DNA to undetectable level (29-31). These drugs are acceptable to most of the patients because they are admitted orally, once daily and without significant side effect. The main problem is HBV DNA tends to relapse in approximately 70% of patients 1-3 years after discontinued therapy (10, 29-31).

When HBV was suppressed by NA therapy, the immune tolerance may also be suppressed. The post treatment relapse is an indirect evidence of losing immune tolerance in such patients (29-31). The post treatment clinical relapse is associated with enhanced Th1 response (35-37). T regulatory (Treg) cells, macrophages and other unidentified factors may play important roles on HBV tolerance (19, 38-41). One of an important phenomenon for patients receiving NA therapy is decrease of Treg cells level (42,43). The post treatment relapse of hepatic necroinflammation is an evidence of the restored HBV specific immune response (44,45).

In addition to the relief of immune tolerance, NA may suppress the HBsAg production from free virus, but no effect is expected for those HBsAg produced by integrated HBV genome. These two types of HBsAg may have some differences on protein conformation and behavior (46,47). The vaccine is produced according to free virus. Therefore, when the HBsAg produced by free virus is suppressed by NA to a low level, the vaccine may be recognized as a new antigen. The immune response elicited by the therapeutic vaccine may have a potential on suppression of free virus.

1.3 Combined HBV vaccine and NA therapy in animal study A Woodchuck animal study suggest entecavir therapy followed by Woodchuck surface (WHs) and core (WHc) DNA vaccination 7 weeks later may induce WHc and WHs specific T cell responses. Two of the 6 animals clear Woodchuck surface antigen (WHBsAg) and product anti-WHBs (48). Similar results can be found in HBV transgenic mice model. Hepatitis B surface (HBs) and hepatitis B core (HBc) specific cellular and humoral response was identified after HBc and HBs protein vaccine therapy (49). In a mouse model with sustained HBV viremia after infection with a recombinant adeno-associated virus carrying a replicable HBV genome. Immunization with the conventional HBV vaccine in the presence of aluminum adjuvant failed to elicit an immune response,but vaccination of mice with HBsAg/CpG induced strong antibody production and T-cell responses(50)

1.4 Combined HBV vaccine and NA therapy in liver transplantation Prevention of HBV reinfection is an important issue in chronic hepatitis B received liver transplantation. HBsAg immunoglobulin (HBIG) is the choice of therapy with evident of good protection (51). However, HBIG is quite expensive and long term therapy is needed. Combination of HBV vaccine and NA therapy had been done in patients received liver transplantation. The initial reports were not good (52-54), but recent studies suggest up to 50% patients response to lamivudine and HBV vaccination combination therapy (55,56) after adjusted dose of HBIG. All these studies did not report severe adverse event using lamivudine and HBV vaccine combination therapy.

1.5 Combined HBV vaccine and NA therapy in patients with chronic hepatitis B To increase response rate many HBV vaccines has been developed by increase immune epitope or posttranslation modifications (57,58) Combination of Lamivudine with therapeutic HBsAg DNA vaccination led to the persistence of T-cell responses (59). An HBV therapeutic vaccine clinical trial studies showed a decrease of HBV replication in hepatitis B e antigen (HBeAg) positive patients received HBV vaccine and lamivudine combination therapy (60).

2. Study objectives To understand the efficacy of combining a 3-year NA and Engerix-B therapy in sustained viral suppression.

3. Investigational plan 3.1 Overall study design This trials will examine the efficacy of NA and Engerix-B combination therapy in chronic hepatitis B.

3.2 Study design Arm A-entecavir pretreated group: Case vs. histological control study. Arm B-tenofovir pretreated group: randomized case and control study. 3.3. Therapy 3.3.1 Entecavir 0.5 mg daily for at least 3 years. 3.3.2 Tenofovir 300 mg daily for at least 3 years. 3.3.3 Five doses of Engerix-B 20 ug during the last 6 month of NA therapy in case group.

Both case and control groups will complete a 3-year NA therapy. The vaccination group will receive a course of Engerix-B vaccination. They will be enrolled at the last 6 months of the NA therapy. Engerix-B will be given at the 0,1st ,2nd 3rd and 6th month after the enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. HBeAg negative chronic hepatitis B
2. Has been receiving a 3-year or more than 3 years entecavir or tenofovir therapy and intending to stop the treatment 6 months later.
3. An inform consent will be obtained after well explanation.

Exclusion Criteria:

1. Pregnant woman.
2. Hepatitis C virus, hepatitis D virus or human immunodeficient virus co-infection.
3. Alcoholism
4. Present with malignant tumor, decompensated liver or renal diseases, present with other major medical illness.
5. Liver cirrhosis, child B or C.

Ages: 31 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
HBV DNA levels during followup period | At 48th weeks of followup after completed combination therapy
  1. Non-responder: When HBV DNA levels were greater than 1*100000 cps/mL and persistence to 1 year after stopped combination therapy, or need other therapy before the end point.
  2. Delayed responder: Those patients with transient elevation of HBV DNA shortly after stopped NA therapy and then become normal ALT and HBV DNA lower than 1*100000 cps/mL without other therapy.
  3. Sustained responder:HBV DNA levels were lower than 1*100000 cps/mL and persistence to 1 year after stopped combination therapy
HBV DNA levels during followup period | At 96th weeks of followup after completed combination therapy
  1. Non-responder: When HBV DNA levels were greater than 1*100000 cps/mL and persistence to 2 years after stopped combination therapy, or need other therapy before the end point.
  2. Delayed responder: Those patients with transient elevation of HBV DNA shortly after stopped NA therapy and then become normal ALT and HBV DNA lower than 1*100000 cps/mL without other therapy.
  3. Sustained responder:HBV DNA levels were lower than 1*100000 cps/mL and persistence to 2 years after stopped combination therapy

SECONDARY OUTCOMES:
Alanine aminotransferase (ALT) level during followup period | At 48 th week of followup after completed combination therapy
  ALT level after completed therapy will be grouped into normal serum ALT level, 1-2x upper limit normal (ULN), 2-5x ULN or >5x ULN. ALT relapse is defined as ALT level >2x ULN.
Alanine aminotransferase (ALT) level during followup period | At 96th weeks of followup after completed combination therapy
  ALT level after completed therapy will be grouped into normal serum ALT level, 1-2x upper limit normal (ULN), 2-5x ULN or >5x ULN. ALT relapse is defined as ALT level >2x ULN.
Quantitative HBsAg (qHBsAg) level during followup period | At 48th week of followup after completed combination therapy
  Serum qHBsAg level after completed therapy will be grouped into lower than 150 international unit (IU)/mL, 500 IU/mL, 500-1000 IU/mL and >1000 IU/mL. Those qHBsAg lower than 150 IU/mL is defined as good serological response.
Quantitative HBsAg (qHBsAg) level during followup period | At 96th week of followup after completed combination therapy
  Serum qHBsAg level after completed therapy will be grouped into lower than 150 international unit (IU)/mL, 500 IU/mL, 500-1000 IU/mL and >1000 IU/mL. Those qHBsAg lower than 150 IU/mL is defined as good serological response.

CONTACTS AND LOCATIONS:
Overall Officials: Dar-In Tai, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen CJ, Wang LY, Yu MW. Epidemiology of hepatitis B virus infection in the Asia-Pacific region. J Gastroenterol Hepatol. 2000 May;15 Suppl:E3-6. doi: 10.1046/j.1440-1746.2000.02124.x. PMID 10921373
- [Background] El Khouri M, dos Santos VA. Hepatitis B: epidemiological, immunological, and serological considerations emphasizing mutation. Rev Hosp Clin Fac Med Sao Paulo. 2004 Aug;59(4):216-24. doi: 10.1590/s0041-87812004000400011. Epub 2004 Sep 9. PMID 15361988
- [Background] Tsay PK, Tai DI, Chen YM, Yu CP, Wan SY, Shen YJ, Lin DY. Impact of gender, viral transmission and aging in the prevalence of hepatitis B surface antigen. Chang Gung Med J. 2009 Mar-Apr;32(2):155-64. PMID 19403005
- [Background] Liaw YF, Brunetto MR, Hadziyannis S. The natural history of chronic HBV infection and geographical differences. Antivir Ther. 2010;15 Suppl 3:25-33. doi: 10.3851/IMP1621. PMID 21041901
- [Background] Burk RD, Hwang LY, Ho GY, Shafritz DA, Beasley RP. Outcome of perinatal hepatitis B virus exposure is dependent on maternal virus load. J Infect Dis. 1994 Dec;170(6):1418-23. doi: 10.1093/infdis/170.6.1418. PMID 7995980
- [Background] Beasley RP, Hwang LY, Lin CC, Leu ML, Stevens CE, Szmuness W, Chen KP. Incidence of hepatitis B virus infections in preschool children in Taiwan. J Infect Dis. 1982 Aug;146(2):198-204. doi: 10.1093/infdis/146.2.198. PMID 7108271
- [Background] Beasley RP, Hwang LY, Lin CC, Ko YC, Twu SJ. Incidence of hepatitis among students at a university in Taiwan. Am J Epidemiol. 1983 Feb;117(2):213-22. doi: 10.1093/oxfordjournals.aje.a113532. PMID 6402925
- [Background] Kamatani Y, Wattanapokayakit S, Ochi H, Kawaguchi T, Takahashi A, Hosono N, Kubo M, Tsunoda T, Kamatani N, Kumada H, Puseenam A, Sura T, Daigo Y, Chayama K, Chantratita W, Nakamura Y, Matsuda K. A genome-wide association study identifies variants in the HLA-DP locus associated with chronic hepatitis B in Asians. Nat Genet. 2009 May;41(5):591-5. doi: 10.1038/ng.348. Epub 2009 Apr 6. PMID 19349983
- [Background] Mbarek H, Ochi H, Urabe Y, Kumar V, Kubo M, Hosono N, Takahashi A, Kamatani Y, Miki D, Abe H, Tsunoda T, Kamatani N, Chayama K, Nakamura Y, Matsuda K. A genome-wide association study of chronic hepatitis B identified novel risk locus in a Japanese population. Hum Mol Genet. 2011 Oct 1;20(19):3884-92. doi: 10.1093/hmg/ddr301. Epub 2011 Jul 12. PMID 21750111
- [Background] Chang SW, Fann CS, Su WH, Wang YC, Weng CC, Yu CJ, Hsu CL, Hsieh AR, Chien RN, Chu CM, Tai DI. A genome-wide association study on chronic HBV infection and its clinical progression in male Han-Taiwanese. PLoS One. 2014 Jun 18;9(6):e99724. doi: 10.1371/journal.pone.0099724. eCollection 2014. PMID 24940741
- [Background] Chu CM, Karayiannis P, Fowler MJ, Monjardino J, Liaw YF, Thomas HC. Natural history of chronic hepatitis B virus infection in Taiwan: studies of hepatitis B virus DNA in serum. Hepatology. 1985 May-Jun;5(3):431-4. doi: 10.1002/hep.1840050315. PMID 3997072
- [Background] Bertoletti A, Ferrari C. Innate and adaptive immune responses in chronic hepatitis B virus infections: towards restoration of immune control of viral infection. Gut. 2012 Dec;61(12):1754-64. doi: 10.1136/gutjnl-2011-301073. Epub 2011 Dec 9. PMID 22157327
- [Background] Das A, Maini MK. Innate and adaptive immune responses in hepatitis B virus infection. Dig Dis. 2010;28(1):126-32. doi: 10.1159/000282075. Epub 2010 May 7. PMID 20460900
- [Background] Fisicaro P, Valdatta C, Boni C, Massari M, Mori C, Zerbini A, Orlandini A, Sacchelli L, Missale G, Ferrari C. Early kinetics of innate and adaptive immune responses during hepatitis B virus infection. Gut. 2009 Jul;58(7):974-82. doi: 10.1136/gut.2008.163600. Epub 2009 Feb 6. PMID 19201769
- [Background] Tan AT, Koh S, Goh W, Zhe HY, Gehring AJ, Lim SG, Bertoletti A. A longitudinal analysis of innate and adaptive immune profile during hepatic flares in chronic hepatitis B. J Hepatol. 2010 Mar;52(3):330-9. doi: 10.1016/j.jhep.2009.12.015. Epub 2010 Jan 13. PMID 20137825
- [Background] Kennedy PTF, Sandalova E, Jo J, Gill U, Ushiro-Lumb I, Tan AT, Naik S, Foster GR, Bertoletti A. Preserved T-cell function in children and young adults with immune-tolerant chronic hepatitis B. Gastroenterology. 2012 Sep;143(3):637-645. doi: 10.1053/j.gastro.2012.06.009. Epub 2012 Jun 15. PMID 22710188
- [Background] Koay LB, Feng IC, Sheu MJ, Kuo HT, Lin CY, Chen JJ, Wang SL, Tang LY, Tsai SL. Hepatitis B virus (HBV) core antigen-specific regulatory T cells confer sustained remission to anti-HBV therapy in chronic hepatitis B with acute exacerbation. Hum Immunol. 2011 Sep;72(9):687-98. doi: 10.1016/j.humimm.2010.11.001. Epub 2011 Jan 6. PMID 21215784
- [Background] Sobao Y, Tomiyama H, Sugi K, Tokunaga M, Ueno T, Saito S, Fujiyama S, Morimoto M, Tanaka K, Takiguchi M. The role of hepatitis B virus-specific memory CD8 T cells in the control of viral replication. J Hepatol. 2002 Jan;36(1):105-15. doi: 10.1016/s0168-8278(01)00264-1. PMID 11804672
- [Background] Bertoletti A, Kennedy PT. The immune tolerant phase of chronic HBV infection: new perspectives on an old concept. Cell Mol Immunol. 2015 May;12(3):258-63. doi: 10.1038/cmi.2014.79. Epub 2014 Sep 1. PMID 25176526
- [Background] Tai DI, Lin SM, Sheen IS, Chu CM, Lin DY, Liaw YF. Long-term outcome of hepatitis B e antigen-negative hepatitis B surface antigen carriers in relation to changes of alanine aminotransferase levels over time. Hepatology. 2009 Jun;49(6):1859-67. doi: 10.1002/hep.22878. PMID 19378345
- [Background] Liaw YF, Tai DI, Chu CM, Lin DY, Sheen IS, Chen TJ, Pao CC. Early detection of hepatocellular carcinoma in patients with chronic type B hepatitis. A prospective study. Gastroenterology. 1986 Feb;90(2):263-7. doi: 10.1016/0016-5085(86)90919-4. PMID 2416625
- [Background] Liaw YF, Tai DI, Chen TJ, Chu CM, Huang MJ. Alpha-fetoprotein changes in the course of chronic hepatitis: relation to bridging hepatic necrosis and hepatocellular carcinoma. Liver. 1986 Jun;6(3):133-7. doi: 10.1111/j.1600-0676.1986.tb00279.x. PMID 2427909
- [Background] Liaw YF, Tai DI, Chu CM, Chen TJ. The development of cirrhosis in patients with chronic type B hepatitis: a prospective study. Hepatology. 1988 May-Jun;8(3):493-6. doi: 10.1002/hep.1840080310. PMID 3371868
- [Background] Liaw YF, Leung N, Kao JH, Piratvisuth T, Gane E, Han KH, Guan R, Lau GK, Locarnini S; Chronic Hepatitis B Guideline Working Party of the Asian-Pacific Association for the Study of the Liver. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. Hepatol Int. 2008 Sep;2(3):263-83. doi: 10.1007/s12072-008-9080-3. Epub 2008 May 10. PMID 19669255
- [Background] European Association For The Study Of The Liver. EASL Clinical Practice Guidelines: management of chronic hepatitis B. J Hepatol. 2009 Feb;50(2):227-42. doi: 10.1016/j.jhep.2008.10.001. Epub 2008 Oct 29. No abstract available. PMID 19054588
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Background] Liaw YF, Jia JD, Chan HL, Han KH, Tanwandee T, Chuang WL, Tan DM, Chen XY, Gane E, Piratvisuth T, Chen L, Xie Q, Sung JJ, Wat C, Bernaards C, Cui Y, Marcellin P. Shorter durations and lower doses of peginterferon alfa-2a are associated with inferior hepatitis B e antigen seroconversion rates in hepatitis B virus genotypes B or C. Hepatology. 2011 Nov;54(5):1591-9. doi: 10.1002/hep.24555. PMID 22045673
- [Background] Marcellin P, Bonino F, Lau GK, Farci P, Yurdaydin C, Piratvisuth T, Jin R, Gurel S, Lu ZM, Wu J, Popescu M, Hadziyannis S; Peginterferon alfa-2a in HBeAg-negative Chronic Hepatitis B Study Group. Sustained response of hepatitis B e antigen-negative patients 3 years after treatment with peginterferon alpha-2a. Gastroenterology. 2009 Jun;136(7):2169-2179.e1-4. doi: 10.1053/j.gastro.2009.03.006. Epub 2009 Mar 19. PMID 19303414
- [Background] Kim YJ, Kim K, Hwang SH, Kim SS, Lee D, Cheong JY, Cho SW. Durability after discontinuation of nucleos(t)ide therapy in chronic HBeAg negative hepatitis patients. Clin Mol Hepatol. 2013 Sep;19(3):300-4. doi: 10.3350/cmh.2013.19.3.300. Epub 2013 Sep 30. PMID 24133668
- [Background] Reijnders JG, Perquin MJ, Zhang N, Hansen BE, Janssen HL. Nucleos(t)ide analogues only induce temporary hepatitis B e antigen seroconversion in most patients with chronic hepatitis B. Gastroenterology. 2010 Aug;139(2):491-8. doi: 10.1053/j.gastro.2010.03.059. Epub 2010 Apr 8. PMID 20381492
- [Background] Jeng WJ, Sheen IS, Chen YC, Hsu CW, Chien RN, Chu CM, Liaw YF. Off-therapy durability of response to entecavir therapy in hepatitis B e antigen-negative chronic hepatitis B patients. Hepatology. 2013 Dec;58(6):1888-96. doi: 10.1002/hep.26549. Epub 2013 Oct 17. PMID 23744454
- [Background] Levrero M, Pollicino T, Petersen J, Belloni L, Raimondo G, Dandri M. Control of cccDNA function in hepatitis B virus infection. J Hepatol. 2009 Sep;51(3):581-92. doi: 10.1016/j.jhep.2009.05.022. Epub 2009 Jun 10. PMID 19616338
- [Background] Zoulim F, Durantel D, Deny P. Management and prevention of drug resistance in chronic hepatitis B. Liver Int. 2009 Jan;29 Suppl 1:108-15. doi: 10.1111/j.1478-3231.2008.01939.x. PMID 19207973
- [Background] Liaw YF. Natural history of chronic hepatitis B virus infection and long-term outcome under treatment. Liver Int. 2009 Jan;29 Suppl 1:100-7. doi: 10.1111/j.1478-3231.2008.01941.x. PMID 19207972
- [Background] Tjwa ET, van Oord GW, Hegmans JP, Janssen HL, Woltman AM. Viral load reduction improves activation and function of natural killer cells in patients with chronic hepatitis B. J Hepatol. 2011 Feb;54(2):209-18. doi: 10.1016/j.jhep.2010.07.009. Epub 2010 Sep 6. PMID 21095036
- [Background] Boni C, Penna A, Bertoletti A, Lamonaca V, Rapti I, Missale G, Pilli M, Urbani S, Cavalli A, Cerioni S, Panebianco R, Jenkins J, Ferrari C. Transient restoration of anti-viral T cell responses induced by lamivudine therapy in chronic hepatitis B. J Hepatol. 2003 Oct;39(4):595-605. doi: 10.1016/s0168-8278(03)00292-7. PMID 12971971
- [Background] Boni C, Penna A, Ogg GS, Bertoletti A, Pilli M, Cavallo C, Cavalli A, Urbani S, Boehme R, Panebianco R, Fiaccadori F, Ferrari C. Lamivudine treatment can overcome cytotoxic T-cell hyporesponsiveness in chronic hepatitis B: new perspectives for immune therapy. Hepatology. 2001 Apr;33(4):963-71. doi: 10.1053/jhep.2001.23045. PMID 11283861
- [Background] Xu L, Yin W, Sun R, Wei H, Tian Z. Liver type I regulatory T cells suppress germinal center formation in HBV-tolerant mice. Proc Natl Acad Sci U S A. 2013 Oct 15;110(42):16993-8. doi: 10.1073/pnas.1306437110. Epub 2013 Oct 2. PMID 24089450
- [Background] Li J, Qiu SJ, She WM, Wang FP, Gao H, Li L, Tu CT, Wang JY, Shen XZ, Jiang W. Significance of the balance between regulatory T (Treg) and T helper 17 (Th17) cells during hepatitis B virus related liver fibrosis. PLoS One. 2012;7(6):e39307. doi: 10.1371/journal.pone.0039307. Epub 2012 Jun 20. PMID 22745730
- [Background] Peng G, Li S, Wu W, Sun Z, Chen Y, Chen Z. Circulating CD4+ CD25+ regulatory T cells correlate with chronic hepatitis B infection. Immunology. 2008 Jan;123(1):57-65. doi: 10.1111/j.1365-2567.2007.02691.x. Epub 2007 Aug 31. PMID 17764450
- [Background] Kondo Y, Kobayashi K, Asabe S, Shiina M, Niitsuma H, Ueno Y, Kobayashi T, Shimosegawa T. Vigorous response of cytotoxic T lymphocytes associated with systemic activation of CD8 T lymphocytes in fulminant hepatitis B. Liver Int. 2004 Dec;24(6):561-7. doi: 10.1111/j.1478-3231.2004.0982.x. PMID 15566505
- [Background] Yu XP, Guo RY, Su ML, Ming DS, Lin CZ, Deng Y, Lin ZZ, Su ZJ. Dynamic Changes of Treg and Th17 Cells and Related Cytokines Closely Correlate With the Virological and Biochemical Response in Chronic Hepatitis B Patients Undergoing Nucleos(t)ide Analogues Treatment. Hepat Mon. 2013 Dec 23;13(12):e15332. doi: 10.5812/hepatmon.15332. eCollection 2013. PMID 24403916
- [Background] Kondo Y, Ueno Y, Kobayashi K, Kakazu E, Shiina M, Inoue J, Tamai K, Wakui Y, Tanaka Y, Ninomiya M, Obara N, Fukushima K, Ishii M, Kobayashi T, Niitsuma H, Kon S, Shimosegawa T. Hepatitis B virus replication could enhance regulatory T cell activity by producing soluble heat shock protein 60 from hepatocytes. J Infect Dis. 2010 Jul 15;202(2):202-13. doi: 10.1086/653496. PMID 20533879
- [Background] Marinos G, Naoumov NV, Williams R. Impact of complete inhibition of viral replication on the cellular immune response in chronic hepatitis B virus infection. Hepatology. 1996 Nov;24(5):991-5. doi: 10.1002/hep.510240503. PMID 8903365
- [Background] Pontesilli O, van Nunen AB, van Riel D, Carotenuto P, Niesters HG, Uytdehaag FG, De Man RA, Osterhaus AD. Hepatitis B virus-specific T cell response in chronic hepatitis B patients treated with lamivudine and interferon-alpha. Liver Int. 2004 Aug;24(4):308-15. doi: 10.1111/j.1478-3231.2004.0922.x. PMID 15287853
- [Background] Freitas N, Cunha C, Menne S, Gudima SO. Envelope proteins derived from naturally integrated hepatitis B virus DNA support assembly and release of infectious hepatitis delta virus particles. J Virol. 2014 May;88(10):5742-54. doi: 10.1128/JVI.00430-14. Epub 2014 Mar 12. PMID 24623409
- [Background] Wang HC, Wu HC, Chen CF, Fausto N, Lei HY, Su IJ. Different types of ground glass hepatocytes in chronic hepatitis B virus infection contain specific pre-S mutants that may induce endoplasmic reticulum stress. Am J Pathol. 2003 Dec;163(6):2441-9. doi: 10.1016/S0002-9440(10)63599-7. PMID 14633616
- [Background] Kosinska AD, Zhang E, Johrden L, Liu J, Seiz PL, Zhang X, Ma Z, Kemper T, Fiedler M, Glebe D, Wildner O, Dittmer U, Lu M, Roggendorf M. Combination of DNA prime--adenovirus boost immunization with entecavir elicits sustained control of chronic hepatitis B in the woodchuck model. PLoS Pathog. 2013;9(6):e1003391. doi: 10.1371/journal.ppat.1003391. Epub 2013 Jun 13. PMID 23785279
- [Background] Buchmann P, Dembek C, Kuklick L, Jager C, Tedjokusumo R, von Freyend MJ, Drebber U, Janowicz Z, Melber K, Protzer U. A novel therapeutic hepatitis B vaccine induces cellular and humoral immune responses and breaks tolerance in hepatitis B virus (HBV) transgenic mice. Vaccine. 2013 Feb 6;31(8):1197-203. doi: 10.1016/j.vaccine.2012.12.074. Epub 2013 Jan 7. PMID 23306359
- [Background] Yang D, Liu L, Zhu D, Peng H, Su L, Fu YX, Zhang L. A mouse model for HBV immunotolerance and immunotherapy. Cell Mol Immunol. 2014 Jan;11(1):71-8. doi: 10.1038/cmi.2013.43. Epub 2013 Sep 30. PMID 24076617
- [Background] Cholongitas E, Goulis J, Akriviadis E, Papatheodoridis GV. Hepatitis B immunoglobulin and/or nucleos(t)ide analogues for prophylaxis against hepatitis b virus recurrence after liver transplantation: a systematic review. Liver Transpl. 2011 Oct;17(10):1176-90. doi: 10.1002/lt.22354. PMID 21656655
- [Background] Di Paolo D, Lenci I, Trinito MO, Carbone M, Longhi C, Tisone G, Angelico M. Extended double-dosage HBV vaccination after liver transplantation is ineffective, in the absence of lamivudine and prior wash-out of human Hepatitis B immunoglobulins. Dig Liver Dis. 2006 Oct;38(10):749-54. doi: 10.1016/j.dld.2006.06.011. Epub 2006 Aug 17. PMID 16916630
- [Background] Lo CM, Liu CL, Chan SC, Lau GK, Fan ST. Failure of hepatitis B vaccination in patients receiving lamivudine prophylaxis after liver transplantation for chronic hepatitis B. J Hepatol. 2005 Aug;43(2):283-7. doi: 10.1016/j.jhep.2005.03.013. PMID 15964658
- [Background] Karasu Z, Ozacar T, Akarca U, Ersoz G, Erensoy S, Gunsar F, Kobat A, Tokat Y, Batur Y. HBV vaccination in liver transplant recipients: not an effective strategy in the prophylaxis of HBV recurrence. J Viral Hepat. 2005 Mar;12(2):212-5. doi: 10.1111/j.1365-2893.2005.00585.x. PMID 15720538
- [Background] Lo CM, Lau GK, Chan SC, Fan ST, Wong J. Efficacy of a pre-S containing vaccine in patients receiving lamivudine prophylaxis after liver transplantation for chronic hepatitis B. Am J Transplant. 2007 Feb;7(2):434-9. doi: 10.1111/j.1600-6143.2006.01636.x. PMID 17283489
- [Background] Di Paolo D, Lenci I, Cerocchi C, Tariciotti L, Monaco A, Brega A, Lotti L, Tisone G, Angelico M. One-year vaccination against hepatitis B virus with a MPL-vaccine in liver transplant patients for HBV-related cirrhosis. Transpl Int. 2010 Nov;23(11):1105-12. doi: 10.1111/j.1432-2277.2010.01104.x. Epub 2010 Aug 19. PMID 20492620
- [Background] Raz R, Koren R, Bass D. Safety and immunogenicity of a new mammalian cell-derived recombinant hepatitis B vaccine containing Pre-S1 and Pre-S2 antigens in adults. Isr Med Assoc J. 2001 May;3(5):328-32. PMID 11411195
- [Background] McDermott AB, Cohen SB, Zuckerman JN, Madrigal JA. Hepatitis B third-generation vaccines: improved response and conventional vaccine non-response--evidence for genetic basis in humans. J Viral Hepat. 1998 Nov;5 Suppl 2:9-11. doi: 10.1046/j.1365-2893.1998.0050s2009.x. PMID 9857354
- [Background] Godon O, Fontaine H, Kahi S, Meritet JF, Scott-Algara D, Pol S, Michel ML, Bourgine M; ANRS HB02 study group. Immunological and antiviral responses after therapeutic DNA immunization in chronic hepatitis B patients efficiently treated by analogues. Mol Ther. 2014 Mar;22(3):675-684. doi: 10.1038/mt.2013.274. Epub 2013 Dec 5. PMID 24394187
- [Background] Hoa PT, Huy NT, Thu le T, Nga CN, Nakao K, Eguchi K, Chi NH, Hoang BH, Hirayama K. Randomized controlled study investigating viral suppression and serological response following pre-S1/pre-S2/S vaccine therapy combined with lamivudine treatment in HBeAg-positive patients with chronic hepatitis B. Antimicrob Agents Chemother. 2009 Dec;53(12):5134-40. doi: 10.1128/AAC.00276-09. Epub 2009 Sep 21. PMID 19770281